CLINICAL TRIAL: NCT06163326
Title: A PHASE 3 RANDOMIZED WITHDRAWAL AND DOSE-UP TITRATION, MULTICENTER EXTENSION STUDY INVESTIGATING THE SAFETY, EFFICACY, AND TOLERABILITY OF RITLECITINIB IN ADULT AND ADOLESCENT PARTICIPANTS WITH NONSEGMENTAL VITILIGO
Brief Title: A 52-Week Study to Learn About the Safety and Effects of Ritlecitinib in Participants With Nonsegmental Vitiligo
Acronym: Tranquillo LTE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B7981041; 2023-505804-42-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Vitiligo
Keywords: Stable vitiligo; Active vitiligo; Adults; Adolescents
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Participants who previously received 1 ritlecitinib 50 mg capsule QD orally from BL to Week 52 in Study B7981040.
  Ritlecitinib 50 mg or Ritlecitinib 100 mg or Placebo will be assigned.
  Interventions: Drug: Ritlecitinib; Drug: Ritlecitinib 100 mg; Drug: Placebo
- Arm 2 (Experimental): Participants who previously received 1 placebo 50 mg capsule QD orally from BL to Week 52 in Study B7981040 Ritlecitinib 50 mg or Ritlecitinib 100 mg or Placebo will be assigned
  Interventions: Drug: Ritlecitinib; Drug: Ritlecitinib 100 mg; Drug: Placebo

INTERVENTIONS:
Drug: Ritlecitinib — Ritlecitinib 50 mg capsule once daily
Drug: Ritlecitinib 100 mg — Ritlecitinib 100 mg capsule once daily
Drug: Placebo — Matching capsule once daily

SUMMARY:
This study is to evaluate how safe and effective ritlecitinib is in participants with non-segmental vitiligo (NSV).

Ritlecitinib is studied in patients with non-segmental vitiligo. Vitiligo is a chronic acquired depigmentation disorder characterized by well-defined pale white patches of skin.

Non-segmental vitiligo is an autoimmune disorder and is the focus of this study. The study will show:

* if the repigmentation (the recovery of pigmentation) achieved in study B7981040 (also called the "parent study") will stay the same or will further increase if you keep receiving the same study medicine (ritlecitinib 50 milligrams or placebo)
* Or if more repigmentation can be achieved if you start receiving ritlecitinib 100 milligrams in this study
* Or how long the repigmentation achieved during the parent study lasts if you start receiving placebo in this study.

This study is seeking for participants who:

* have non-segmental vitiligo (either active or stable) and
* received ritlecitinib or placebo for 52 weeks in the parent study. A placebo looks exactly like the study capsule but does not contain any medicine in it.

All participants in this study will receive the study medicine or placebo. The study medicine (ritlecitinib 50 milligrams or 100 milligrams) or placebo are capsules that are taken by mouth at home every day. On study visit days, you must take the medication at the study site, and not at home.

Participants may receive the study medicine or placebo for up to 52 weeks.

The study will look at the experiences of people receiving the study medicine. This will help see if ritlecitinib is better for treating vitiligo.

Participants will be involved in this study for a maximum of 60 weeks. During this time, they will have 9 study visits during the study.

Ritlecitinib 50 mg is an approved drug for the treatment of severe Alopecia Areata (a disease with similar abnormal changes in the body functions like vitiligo) in the US, EU and Japan. China, Great Britain and other market applications are pending.

ELIGIBILITY:
Inclusion Criteria:

* Participants ≥18 years of age at Screening in Study B7981040. Adolescents (12 to <18 years of age at Screening in the parent study) are also eligible for this study if approved by the local IRB/EC and regulatory health authority.
* Participants who met the eligibility criteria and completed 52 weeks of study intervention for stable or active nonsegmental vitiligo in Study B7981040
* The BL visit/first dose in Study B7981041 must be within 30 days after the week 52 visit in Study B7981040

Exclusion Criteria:

* Participant met the parent study (Study 7981040) discontinuation criteria or discontinued the parent study for any safety-related event
* Any active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2027-04-23 (Estimated); Study Completion 2027-04-23 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), and adverse events (AEs) leading to discontinuation | Screening up to at least 30 days after last dose of study drug (week 52 or Early Termination)
  To evaluate the long-term safety and tolerability of ritlecitinib in adult and adolescent participants with non-segmental vitiligo
Incidence of clinically significant laboratory abnormalities | Screening up to at least 30 days after last dose of study drug (week 52 or Early Termination)
  To evaluate the long-term safety and tolerability of ritlecitinib in adult and adolescent participants with non-segmental vitiligo

SECONDARY OUTCOMES:
Response based on T-VASI75 at weeks 4, 8, 12, 24, 36 and 52 | Baseline to week 52
  Proportion of participants achieving at least a 75% improvement in T-VASI from Baseline
Response based on F-VASI75 at weeks 4, 8, 12, 24, 36 and 52 | Baseline to week 52
  Proportion of participants achieving at least a 75% improvement in F-VASI from Baseline
Response based on T-VASI50 at weeks 4, 8, 12, 24, 36 and 52 | Baseline to Week 52
  Proportion of participants achieving at least a 50% improvement in T-VASI from Baseline
Response based on F-VASI50 at weeks 4, 8, 12, 24, 36 and 52 | Baseline to week 52
  Proportion of participants achieving at least a 50% improvement in F-VASI from Baseline
Response based on T-VASI90 at weeks 4, 8, 12, 24, 36 and 52 | Baseline to week 52
  Proportion of participants achieving at least a 90% improvement in T-VASI from Baseline
Response based on F-VASI90 at weeks 4, 8, 12, 24, 36 and 52 | Baseline to week 52
  Proportion of participants achieving at least a 90% improvement in F-VASI from Baseline
Response based on T-VASI100 at weeks 4, 8, 12, 24, 36 and 52 | Baseline to week 52
  Proportion of participants achieving at least a 100% improvement in T-VASI from Baseline
Response based on F-VASI100 at weeks 4, 8, 12, 24, 36 and 52 | Baseline to week 52
  Proportion of participants achieving at least a 100% improvement in F-VASI from Baseline
Patient Global Impression of Severity-Face (PGIS-F) at weeks 24, 36, and 52 | Baseline to week 52
  To assess the effect of ritlecitinib compared to placebo on the PGIC-F at weeks 24, 36, and 52
Patient Global Impression of Severity-Overall Vitiligo (PGIS-V) at weeks 24, 36, and 52 | Baseline to week 52
  To assess the effect of ritlecitinib compared to placebo on the PGIC-V at Week 24, 36, and 52
Patient Global Impression of Change-Face (PGIC-F) at week 24, 36, and 52 | Baseline to week 52
  To assess the effect of ritlecitinib compared to placebo on the PGIC-F at Week 24, 36, and 52
Patient Global Impression of Change- Overall vitiligo (PGIC-V) at weeks 24, 36, and 52 | Baseline to week 52
  To assess the effect of ritlecitinib compared to placebo on the PGIC-V at weeks 24, 36, and 52
Proportion of participants achieving disease stabilization | Baseline to week 52
  The difference in the proportion of participants with stable disease at all scheduled timepoints
Percentage change from baseline (%CFB) in F-VASI at weeks 4, 8, 12, 24, 36, and 52 | Baseline to week 52
  To compare the efficacy of ritlecitinib 100mg QD, 50mg QD, and placebo
Percentage change from baseline (%CFB) in T-VASI at weeks 4, 8, 12, 24, 36, and 52 | Baseline to week 52
  To compare the efficacy of ritlecitinib 100mg QD, 50mg QD, and placebo
Time to loss of response (<F-VASI75 and <T-VASI50 at the same visit). | Baseline to week 52
  To compare the efficacy of ritlecitinib 100 mg QD, 50 mg QD, and placebo

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (74):
- United States (22):
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - Marvel Clinical Research, Huntington Beach, California
  - Wallace Medical Group, Inc, Los Angeles, California
  - Encore Medical Research of Boynton Beach, Boynton Beach, Florida
  - Skin Care Research, Hollywood, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - DelRicht Research, Baton Rouge, Louisiana
  - Lawrence J. Green, MD LLC, Rockville, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - SUNY Downstate Health Sciences University, Brooklyn, New York
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - Clinical & Translational Research Center (CTRC), Chapel Hill, North Carolina
  - Accellacare - Wilmington, Wilmington, North Carolina
  - Wilmington Health, PLLC, Wilmington, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Remington-Davis, Inc, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Modern Research Associates, PLLC, Dallas, Texas
  - Alpesh D. Desai, DO PLLC, Houston, Texas
  - Austin Institute for Clinical Research, Houston, Texas
- Australia (5):
  - The Skin Hospital, Darlinghurst, New South Wales
  - North Eastern Health Specialists, Campbelltown, South Australia
  - Skin Health Institute Inc., Carlton, Victoria
  - Dr Rodney Sinclair Pty Ltd, East Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Bulgaria (3):
  - Medical Centre "Asklepiy", Dupnitsa, Kyustendil
  - Diagnostic Consultative Center Aleksandrovska, Sofia, Sofia (stolitsa)
  - UMHAT "Prof. Dr. Stoyan Kirkovich"AD, Stara Zagora
- Canada (7):
  - Dermatology Research Institute, Calgary, Alberta
  - CaRe Clinic, Red Deer, Alberta
  - Lynderm Research Inc., Markham, Ontario
  - DermEdge Research, Mississauga, Ontario
  - North York Research Inc, Toronto, Ontario
  - Centre de Recherche Dermatologique du Quebec metropolitain, Québec
  - Centre de Recherche Saint-Louis inc., Québec
- China (6):
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - The First Hospital of Wuhan, Wuhan, Hubei
  - The First Hospital of China Medical University/Dermatology and STD Department, Shenyang, Liaoning
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
- Germany (3):
  - Praxis Leitz und Kollegen, Stuttgart, Baden-Wurttemberg
  - Fachklinik Bad Bentheim, Bad Bentheim, Lower Saxony
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
- Japan (6):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Tohoku University Hospital, Sendai, Miyagi
  - Dermatology and Ophthalmology Kume Clinic, Sakai, Osaka
  - Nippon Medical School Hospital, Bunkyo-ku, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo
  - Yamanashi Prefectural Central Hospital, Kofu, Yamanashi
- Mexico (4):
  - Hospital Infantil de Mexico Federico Gomez, Mexico City, Mexico City
  - Centro de Dermatologia de Monterrey, Monterrey, Nuevo León
  - Arké SMO S.A de C.V, Veracruz
  - Sociedad de Metabolismo y Corazon S.C., Veracruz
- Poland (5):
  - DermoDent Centrum Medyczne Aldona Czajkowska Rafał Czajkowski s.c., Osielsko, Kuyavian-Pomeranian Voivodeship
  - Royalderm Agnieszka Nawrocka, Warsaw, Masovian Voivodeship
  - Twoja Przychodnia SCM, Szczecin, West Pomeranian Voivodeship
  - Dermoklinika - Centrum Medyczne spółka cywilna M. Kierstan, J. Narbutt, A. Lesiak, Lodz, Łódź Voivodeship
  - Dermedic Jacek Zdybski, Ostrowiec Świętokrzyski, Świętokrzyskie Voivodeship
- South Korea (3):
  - The Catholic University Of Korea St. Vincent's Hospital, Suwon, Kyǒnggi-do
  - Ajou University Hospital, Suwon, Kyǒnggi-do
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [seoul]
- Spain (5):
  - Hospital Universitario Reina Sofia, Córdoba, Andalusia
  - Hospital Clínic de Barcelona, Barcelona, Catalunya [cataluña]
  - Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas de Gran Canaria, LAS Palmas
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid, Comunidad de
  - AUDIKA, Córdoba
- Turkey (Türkiye) (4):
  - Istanbul Universitesi Cerrahpasa, Istanbul- Fatih, Istanbul
  - Marmara Universitesi Pendik Egitim Arastirma Hastanesi, Istanbul, İ̇stanbul
  - Erciyes Universitesi Tıp Fakultesi Hastaneleri, Kayseri
  - Celal Bayar University Hafsa Sultan Hospital, Manisa
- Guy's & St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7981041